CLINICAL TRIAL: NCT06868940
Title: Clinical Application Study of Wearable Multi-channel Electrocardiogram Acquisition Equipment in the Diagnosis of Myocardial Ischemia in Patients with Suspected Coronary Heart Disease
Brief Title: Clinical Application Study of Wearable Multi-channel Electrocardiogram Acquisition Equipment in the Diagnosis of Myocardial Ischemia in Patients with Suspected CHD
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Sichuan University
Other Study IDs: WestChinaH-CVD-008
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Coronary Arterial Disease (CAD); Myocardial Ischaemia; Wearable Electronic Devices
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: wearable multi-channel ECG acquisition devices — If patients do not meet the exclusion criteria, they will wear the wearable multi-channel ECG device for 7 days after enrollment, followed by a myocardial SPECT examination; there is no specific order for these examinations. After enrollment, baseline information of the patients (such as age, gender, height, weight, etc.), comorbidities (such as hypertension, diabetes, hyperlipidemia, chronic kidney disease, etc.), and auxiliary examination data (such as complete blood count, biochemistry, cardiac injury markers, BNP, echocardiography, wearable multi-channel ECG device data, SPECT-related examination data, such as ST-segment, total load score, total rest score, etc.) will be collected. The endpoint of this study is to evaluate the sensitivity, specificity, and accuracy of the wearable multi-channel ECG device in assessing myocardial ischemia in CHD.

SUMMARY:
Backgroud: With the widespread application of artificial intelligence, sensor technology, and wearable technology in clinical and daily life, wearable devices have shown a promising application prospect and tremendous potential. Currently, both domestic and international clinical applications of wearable ECG devices for the diagnosis and treatment of coronary heart disease are mostly single-lead ECG wearable devices or simulated multi-lead wearable ECG monitoring devices, which are widely used in the diagnosis of arrhythmias such as atrial fibrillation. There is a lack of clinical diagnostic efficacy research on myocardial ischemia in coronary heart disease.

Aim: To investigate the diagnostic efficacy of wearable multi-channel ECG acquisition devices for myocardial ischemia in suspected CHD patients Methods：Assessing the sensitivity, specificity, and accuracy of wearable multi-channel ECG devices in diagnosing myocardial ischemia in coronary heart disease by comparing with the "gold standard" SPECT-MPI.The target recruitment is 107 suspected coronary heart disease myocardial ischemia patients.If patients do not meet the exclusion criteria, they will wear the wearable multi-channel ECG device for 7 days after enrollment, followed by a myocardial SPECT examination; there is no specific order for these examinations. After enrollment, baseline information of the patients (such as age, gender, height, weight, etc.), comorbidities (such as hypertension, diabetes, hyperlipidemia, chronic kidney disease, etc.), and auxiliary examination data (such as complete blood count, biochemistry, cardiac injury markers, BNP, echocardiography, wearable multi-channel ECG device data, SPECT-related examination data, such as ST-segment, total load score, total rest score, etc.) will be collected. The endpoint of this study is to evaluate the sensitivity, specificity, and accuracy of the wearable multi-channel ECG device in assessing myocardial ischemia in CHD.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a participant must meet all of the following criteria:

  1. Age > 18 years old;
  2. Patients suspected of having coronary heart disease with myocardial ischemia;
  3. Capable of using wearable ECG monitoring devices properly;
  4. Informed consent obtained from the patient.

Exclusion Criteria:

* If a patient meets any of the following conditions, they will be excluded:

  1. Hemodynamic instability;
  2. Second to third-degree atrioventricular block, sustained ventricular tachycardia, ventricular fibrillation, severe sinus bradycardia (heart rate < 40 beats/min).
  3. Known congenital heart disease, severe valvular heart disease, acute heart failure, and decompensated chronic heart failure;
  4. Severe comorbidities: Other diseases expected to have a life expectancy of ≤12 months; bronchial asthma or severe liver and kidney dysfunction; history of severe renal or liver function abnormalities (glomerular filtration rate < 30 ml/(min·1.73²m²), liver failure, cirrhosis, portal hypertension, or active hepatitis), neutropenia, thrombocytopenia;
  5. Allergy to adenosine;
  6. Imaging failure, such as patient movement during the acquisition process or too rapid injection of the imaging agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of having coronary heart disease with myocardial ischemia may exhibit symptoms such as angina, myocardial infarction, arrhythmias, heart failure, and sudden death. They may show signs of myocardial ischemia on an electrocardiogram, such as changes in the ST segment or T wave, but these changes are not specific and require further examination for confirmation.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and accuracy | After enrollment, wear the wearable multi-channel ECG device for 7 days, followed by the completion of a myocardial SPECT examination.
  Sensitivity, specificity, and accuracy of wearable multi-channel ECG acquisition devices in diagnosing myocardial ischemia in coronary heart disease.